CLINICAL TRIAL: NCT03946449
Title: A Pilot Open Label, Multi-dose, Phase 2 Study to Assess the Safety and Efficacy of Fazirsiran (TAK-999, ARO-AAT) in Patients With Alpha-1 Antitrypsin Deficiency Associated Liver Disease (AATD)
Brief Title: Study of Fazirsiran (TAK-999, ARO-AAT) in Patients With Alpha-1 Antitrypsin Deficiency Associated Liver Disease (AATD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AROAAT2002; 2019-000068-86 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ARO-AAT 100 mg Cohort 1b (Experimental): Primary Study Period (6-12 months): 100 mg dose of subcutaneous ARO-AAT for a minimum of 3 doses, with 2 optional treatment extension periods. Treatment Extension I (12 months): 100 mg dose of subcutaneous AROAAT every 12 weeks (Q12W). Treatment Extension II (up to 24 Months): 100 mg dose of subcutaneous ARO-AAT Q12W.
  Interventions: Drug: ARO-AAT
- ARO-AAT 200 mg Cohort 1 (Experimental): Primary Study Period (6-12 months): 200 mg dose of subcutaneous ARO-AAT for a minimum of 3 doses, with 2 optional treatment extension periods. Treatment Extension I (12 months): 200 mg dose of subcutaneous AROAAT Q12W. Treatment Extension II (up to 24 Months): 200 mg dose of subcutaneous ARO-AAT Q12W.
  Interventions: Drug: ARO-AAT
- ARO-AAT 200 mg Cohort 2 (Experimental): Primary Study Period (6-12 months): 200 mg dose of subcutaneous ARO-AAT for a minimum of 5 doses, with optional treatment extension periods. Treatment Extension I (12 months): 200 mg dose of subcutaneous AROAAT Q12W. Treatment Extension II (up to 24 Months): 200 mg dose of subcutaneous ARO-AAT Q12W.
  Interventions: Drug: ARO-AAT

INTERVENTIONS:
Drug: ARO-AAT — solution for subcutaneous injection
  Other Names: Fazirsiran Injection; TAK-999

SUMMARY:
The purpose of this study is to evaluate the the safety and efficacy of the investigational product, fazirsiran (TAK-999, ARO-AAT), administered subcutaneously to patients with alpha-1 antitrypsin deficiency associated liver disease (AATD).

DETAILED DESCRIPTION:
Participants will be enrolled to receive multiple subcutaneous injections of fazirsiran (TAK-999, ARO-AAT). All eligible participants will require a pre-dose biopsy completed as part of the study within the screening window. All participants will undergo an end of study (EOS) biopsy. Treated participants will be offered the opportunity to continue treatment in an open label extension during which they will undergo a final biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AATD
* Liver biopsy indicating Metavir F1-F3 liver fibrosis based on local pathology read.
* Women of childbearing potential must have a negative pregnancy test, cannot be breast feeding, and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements
* Non-smoker for at least 1 year
* No abnormal finding of clinical relevance at screening

Exclusion Criteria:

* Clinically significant health concerns other than AATD
* Previous diagnosis or diagnosis at Screening of definitive liver cirrhosis
* Regular use of alcohol within one month prior to Screening
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study involving therapeutic intervention
* Use of illicit drugs within 1 year prior to Screening

Note: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Research Center 1, Vienna, Austria
- Research Center 1, Aachen, Germany
- United Kingdom (2):
  - Research Center 3, Cambridge
  - Research Center 2, Edinburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strnad P, Mandorfer M, Choudhury G, Griffiths W, Trautwein C, Loomba R, Schluep T, Chang T, Yi M, Given BD, Hamilton JC, San Martin J, Teckman JH. Fazirsiran for Liver Disease Associated with Alpha1-Antitrypsin Deficiency. N Engl J Med. 2022 Aug 11;387(6):514-524. doi: 10.1056/NEJMoa2205416. Epub 2022 Jun 25. PMID 35748699

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All eligible subjects required a pre-dose biopsy completed as part of the study within the screening window. Participants consisted of male and female adult homozygous Z allele individuals (PiZZ; based on genotype completed at Screening or from a source verifiable document) alpha-1 antitrypsin patients.
Groups:
- ARO-AAT 100 mg Cohort 1b: Primary Study Period (6-12 months): 100 mg dose of subcutaneous ARO-AAT for a minimum of 3 doses, with 2 optional treatment extension periods. Treatment Extension I (12 months): 100 mg dose of subcutaneous ARO-AAT every 12 weeks (Q12W). Treatment Extension II (up to 24 Months): 100 mg dose of subcutaneous ARO-AAT Q12W. As of global protocol version 7.0 (21-Jul-2022) / German protocol version 2.6 (29-Jul-2022) and after applicable regulatory, Ethics Committee and local approval, participants in Cohort 1b switched from 100 mg to 200 mg while maintaining their dosing schedule.
  The maximum number of doses for participants completing the treatment extension periods was 15 doses.
- ARO-AAT 200 mg Cohort 1: Primary Study Period (6-12 months): 200 mg dose of subcutaneous ARO-AAT for a minimum of 3 doses, with 2 optional treatment extension periods. Treatment Extension I (12 months): 200 mg dose of subcutaneous ARO-AAT Q12W. Treatment Extension II (up to 24 Months): 200 mg dose of subcutaneous ARO-AAT Q12W.
  The maximum number of doses for participants completing the treatment extension periods was 15 doses.
- ARO-AAT 200 mg Cohort 2: Primary Study Period (6-12 months): 200 mg dose of subcutaneous ARO-AAT for a minimum of 5 doses, with optional treatment extension periods. Treatment Extension I (12 months): 200 mg dose of subcutaneous ARO-AAT Q12W. Treatment Extension II (up to 24 months): 200 mg dose of subcutaneous ARO-AAT Q12W.
  The maximum number of doses for participants completing the treatment extension periods was 17 doses.
Period: Primary Study Period
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1 | ARO-AAT 200 mg Cohort 2
Started | 4 | 4 | 8
Completed | 4 | 4 | 8
Not Completed | 0 | 0 | 0
Period: Treatment Extension I
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1 | ARO-AAT 200 mg Cohort 2
Started | 4 | 4 | 7 (1 participant completed the primary study period, but did not continue in the treatment extension period.)
Completed | 4 | 4 | 7
Not Completed | 0 | 0 | 0
Period: Treatment Extension II
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1 | ARO-AAT 200 mg Cohort 2
Started | 4 | 4 | 7
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 3
Not completed — Rolled over to another study | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1 | ARO-AAT 200 mg Cohort 2 | Total
Number analyzed (Participants) | 4 | 4 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.01) | 44.5 (17.00) | 54.6 (13.68) | 52.1 (14.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 3 | 4 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 8 | 16
Insoluble Z-Alpha 1 Antitrypsin (Z-AAT) [Mean (Standard Deviation); unit: nmol/g] | 35.9750 (16.51694) | 33.2750 (53.31019) | 37.4500 (27.73075) | 36.0375 (31.38345)
Soluble Z-AAT [Mean (Standard Deviation); unit: nmol/g] | 26.3500 (5.18813) | 24.3000 (10.58899) | 23.3125 (7.59914) | 24.3188 (7.50984)
Total Z-AAT [Mean (Standard Deviation); unit: nmol/g] | 62.3250 (15.81210) | 57.5750 (59.65391) | 60.7625 (34.04199) | 60.3563 (36.13456)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Liver Z-AAT, Insoluble Liver-ZAAT, and Soluble Liver Z-AAT at Week 24: Cohorts 1/1b
Time Frame: Baseline, Week 24
Population: Full Analysis Set: all participants who received at least one dose of study drug and had baseline and post-dose liver biopsy histology results available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
percent change
  Total Liver Z-AAT | -83.07 (5.830) | -79.84 (10.519)
  Insoluble Liver-ZAAT | -81.58 (6.947) | -12.91 (131.702)
  Soluble Liver Z-AAT | -85.36 (4.835) | -88.18 (5.718)

2. Primary Outcome: Percent Change From Baseline in Total Liver Z-AAT, Insoluble Liver-ZAAT, and Soluble Liver Z-AAT at Week 48: Cohort 2
Time Frame: Baseline, Week 48
Population: Full Analysis Set: all participants who received at least one dose of study drug and had baseline and post-dose liver biopsy histology results available. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 7
percent change
  Total Liver Z-AAT | -90.26 (9.029)
  Insoluble Liver-ZAAT | -84.83 (19.920)
  Soluble Liver Z-AAT | -92.64 (7.482)

3. Secondary Outcome: Percent Change From Baseline in Serum Z-AAT Over Time: Cohorts 1/1b
Time Frame: Baseline, Weeks 2, 4, 6, 16, 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
percent change
  Week 2 | -69.12 (12.381) | -77.28 (7.394)
  Week 4 | -80.24 (8.880) | -88.07 (4.931)
  Week 6 | -87.27 (6.140) | -91.79 (3.795)
  Week 16 | -78.61 (9.186) | -83.08 (6.269)
  Week 24 | -83.85 (5.426) | -89.47 (3.738)

4. Secondary Outcome: Percent Change From Baseline in Serum Z-AAT Over Time: Cohort 2
Time Frame: Baseline, Weeks 2, 4, 6, 16, 22, 28, 34, 40, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
percent change
  Week 2 | -72.08 (8.645)
  Week 4 | -82.22 (7.476)
  Week 6 | -89.92 (4.024)
  Week 16 | -85.76 (6.106)
  Week 22 | -90.87 (4.246)
  Week 28 | -85.06 (7.847)
  Week 34 | -89.54 (5.434)
  Week 40 | -84.12 (12.433)
  Week 48 | -89.58 (5.419)

5. Secondary Outcome: Alanine Aminotransferase (ALT) Values Over Time: Cohorts 1/1b
Time Frame: Baseline (Day 1), Day 2, Week 2, Week 4, Week 4 (24-48h post dose), Week 6, Week 16, Week 16 (24/48h post dose), Week 24
Population: Safety Analysis Set: all participants who received at least one dose of study drug. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
U/L
  Baseline (Day 1) | 58.5 (41.36) | 87.8 (30.42)
  Day 2 (24-48 hr post-dose) | 58.5 (42.68) | 88.3 (32.72)
  Week 2 | 76.5 (55.24) | 99.8 (53.89)
  Week 4 | 62.3 (35.77) | 106.5 (42.57)
  Week 4 (24-48 hr post-dose) | 60.3 (33.97) | 99.0 (38.58)
  Week 6 | 49.8 (25.16) | 77.0 (20.85)
  Week 16: number analyzed (Participants) | 3 | 4
  Week 16 | 35.7 (8.50) | 49.8 (5.25)
  Week 16 (24-48 hr post-dose): number analyzed (Participants) | 4 | 3
  Week 16 (24-48 hr post-dose) | 31.5 (8.85) | 42.7 (3.06)
  Week 24 | 27.8 (9.29) | 39.5 (3.11)

6. Secondary Outcome: ALT Values Over Time: Cohort 2
Time Frame: Baseline (Day 1), Day 2, Week 2, Week 4, Week 4 (24-48h post dose), Week 6, Week 16, Week 16 (24/48h post dose), Week 22, Week 28, Week 34, Week 40, Week 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
U/L
  Baseline (Day 1) | 62.1 (14.98)
  Day 2 (24-48 hr post-dose) | 58.6 (15.59)
  Week 2: number analyzed (Participants) | 7
  Week 2 | 61.9 (20.17)
  Week 4 | 55.3 (14.09)
  Week 4 (24-48 hr post-dose) | 53.0 (14.83)
  Week 6: number analyzed (Participants) | 7
  Week 6 | 54.9 (9.79)
  Week 16 | 39.6 (13.13)
  Week 16 (24-48 hr post-dose) | 37.5 (11.61)
  Week 22 | 41.0 (14.58)
  Week 28: number analyzed (Participants) | 7
  Week 28 | 36.7 (15.76)
  Week 34 | 39.4 (11.13)
  Week 40 | 33.4 (10.08)
  Week 48: number analyzed (Participants) | 6
  Week 48 | 34.5 (10.54)

7. Secondary Outcome: Gamma Glutamyl Transferase (GGT) Values Over Time: Cohorts 1/1b
Time Frame: as for outcome 5
Population: Safety Analysis Set: all participants who received at least one dose of study drug; n=participants with an assessment at given time point. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
U/L
  Baseline (Day 1) | 70.8 (35.30) | 244.8 (355.68)
  Day 2 (24-48 hr post-dose) | 70.5 (39.07) | 247.3 (358.01)
  Week 2 | 66.0 (37.15) | 210.8 (304.4)
  Week 4 | 73.0 (43.37) | 222.0 (334.85)
  Week 4 (24-48 hr post-dose) | 70.0 (45.19) | 210.3 (312.0)
  Week 6 | 64.0 (35.62) | 199.3 (292.28)
  Week 16 | 48.0 (23.25) | 135.3 (190.31)
  Week 16 (24-48 hr post-dose): number analyzed (Participants) | 4 | 3
  Week 16 (24-48 hr post-dose) | 48.0 (22.38) | 161.7 (212.17)
  Week 24 | 52.3 (28.31) | 112.0 (156.92)

8. Secondary Outcome: GGT Values Over Time: Cohort 2
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
U/L
  Baseline (Day 1) | 62.5 (31.09)
  Day 2 (24-48 hr post-dose) | 62.1 (33.21)
  Week 2: number analyzed (Participants) | 7
  Week 2 | 60.6 (33.14)
  Week 4 | 59.1 (49.82)
  Week 4 (24-48 hr post-dose) | 57.6 (46.91)
  Week 6: number analyzed (Participants) | 7
  Week 6 | 58.0 (36.21)
  Week 16 | 49.1 (36.84)
  Week 16 (24-48 hr post-dose) | 48.3 (38.68)
  Week 22 | 48.5 (34.85)
  Week 28 | 44.5 (34.62)
  Week 34 | 45.3 (31.37)
  Week 40 | 45.3 (38.20)
  Week 48 | 48.5 (45.05)

9. Secondary Outcome: Fibrosis-4 Index (FIB4) Score Values Over Time: Cohorts 1/1b
Description: The FIB 4 score evaluates the degree of fibrosis in patients suspected of or already diagnosed with hepatic fibrosis. FIB-4 is calculated as (Age (years) * aspartate aminotransferase) / (platelets * √(ALT)).
  The result provided from the above equation is interpreted according to 2 cut off values: FIB 4 <1.45 indicates absence of cirrhosis (with a negative predictive value of 90% for advanced fibrosis); FIB 4 between 1.45 - 3.25 are deemed inconclusive; FIB 4 >3.25 indicates cirrhosis (with a positive predictive value of 65% for advanced fibrosis).
Time Frame: Baseline (Day 1), Day 2 (24-48 hr post-dose), Week 2, Week 4, Week 4 (24-48 hr post-dose), Week 6, Week 16, Week 16 (24-48 hr post-dose), Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: numerical score
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
numerical score
  Baseline (Day 1) | 1.425 (0.3613) | 1.583 (0.9085)
  Day 2 (24-48 hr post-dose) | 1.353 (0.2699) | 1.618 (0.9668)
  Week 2 | 1.580 (0.5806) | 1.900 (1.3056)
  Week 4 | 1.260 (0.3840) | 1.750 (1.3273)
  Week 4 (24-48 hr post-dose) | 1.333 (0.4194) | 1.760 (1.3867)
  Week 6 | 1.355 (0.4612) | 2.013 (1.1073)
  Week 16: number analyzed (Participants) | 3 | 4
  Week 16 | 1.257 (0.3326) | 1.605 (1.221)
  Week 16 (24-48 hr post-dose): number analyzed (Participants) | 3 | 3
  Week 16 (24-48 hr post-dose) | 1.227 (0.2230) | 1.940 (1.6210)
  Week 24 | 1.265 (0.3196) | 1.688 (1.2563)

10. Secondary Outcome: FIB4 Score Values Over Time: Cohort 2
Description: as for outcome 9
Time Frame: Baseline (Day 1), Day 2 (24-48 hr post-dose), Week 2, Week 4, Week 4 (24-48 hr post-dose), Week 6, Week 16, Week 16 (24-48 hr post-dose), Week 22, Week 28, Week 28 + 1 day, Week 34, Week 40, Week 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: numerical score
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
numerical score
  Baseline (Day 1) | 1.395 (0.6634)
  Day 2 (24-48 hr post-dose) | 1.543 (0.8209)
  Week 2: number analyzed (Participants) | 7
  Week 2 | 1.383 (0.6358)
  Week 4 | 1.420 (0.7054)
  Week 4 (24-48 hr post-dose) | 1.356 (0.6344)
  Week 6: number analyzed (Participants) | 7
  Week 6 | 1.367 (0.6419)
  Week 16 | 1.299 (0.5636)
  Week 16 (24-48 hr post-dose) | 1.271 (0.6521)
  Week 22 | 1.336 (0.6269)
  Week 28: number analyzed (Participants) | 7
  Week 28 | 1.377 (0.7152)
  Week 34: number analyzed (Participants) | 7
  Week 34 | 1.239 (0.7527)
  Week 40 | 1.319 (0.5782)
  Week 48: number analyzed (Participants) | 5
  Week 48 | 1.502 (0.7680)

11. Secondary Outcome: Aspartate Aminotransferase-to-platelet Ratio Index (APRI) Values Over Time: Cohorts 1/1b
Description: The APRI suggests the level of hepatic fibrosis and possible liver disease. APRI is calculated as 100*(aspartate aminotransferase/40) / platelets. Scores indicate the following: < 0.5 = fibrosis is ruled out; 0.5 - 0.7 = associated with some kind of liver damage; 0.7 - 1 = significant fibrosis; > 1 = associated with cirrhosis.
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: numerical score
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
numerical score
  Baseline (Day 1) | 0.485 (0.2249) | 0.745 (0.3877)
  Day 2 (24-48 hr post-dose) | 0.463 (0.2133) | 0.753 (0.3923)
  Week 2 | 0.633 (0.3349) | 0.910 (0.5231)
  Week 4 | 0.463 (0.2185) | 0.810 (0.4031)
  Week 4 (24-48 hr post-dose) | 0.468 (0.1921) | 0.785 (0.4171)
  Week 6 | 0.433 (0.1688) | 0.918 (0.1834)
  Week 16 | 0.343 (0.0404) | 0.555 (0.3008)
  Week 16 (24-48 hr post-dose) | 0.330 (0.0700) | 0.603 (0.4203)
  Week 24 | 0.310 (0.0970) | 0.513 (0.2892)

12. Secondary Outcome: APRI Values Over Time: Cohort 2
Description: as for outcome 11
Time Frame: Baseline (Day 1), Day 2 (24-48 hr post-dose), Week 2, Week 4, Week 4 (24-48 hr post-dose), Week 6, Week 16, Week 16 (24-48 hr post-dose), Week 22, Week 28, Week 34, Week 40, Week 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: numerical score
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
numerical score
  Baseline (Day 1) | 0.500 (0.2102)
  Day 2 (24-48 hr post-dose) | 0.515 (0.2023)
  Week 2: number analyzed (Participants) | 7
  Week 2 | 0.486 (0.1551)
  Week 4 | 0.479 (0.2226)
  Week 4 (24-48 hr post-dose) | 0.454 (0.2127)
  Week 6: number analyzed (Participants) | 7
  Week 6 | 0.463 (0.1678)
  Week 16 | 0.372 (0.1812)
  Week 16 (24-48 hr post-dose) | 0.358 (0.2160)
  Week 22 | 0.386 (0.2011)
  Week 28: number analyzed (Participants) | 7
  Week 28 | 0.387 (0.2642)
  Week 34: number analyzed (Participants) | 7
  Week 34 | 0.379 (0.2449)
  Week 40 | 0.349 (0.1768)
  Week 48: number analyzed (Participants) | 5
  Week 48 | 0.440 (0.2310)

13. Secondary Outcome: N-Terminal Type III Collagen Propeptide (PRO-C3) Values Over Time: Cohorts 1/1b
Description: PRO-C3 may be a biomarker for the formation of fibrotic tissue in the liver. For serum, the normal range is 6.1 - 13.8 ng/mL (based on a study of human serum samples from healthy men and women). Due to ethnic, dietary and age variations, the reference limits given may not apply to all populations. A reduction in Pro-C3 over time may indicate a reduction in hepatic fibrogenesis.
Time Frame: Baseline, Weeks 4, 16, 24
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
μg/L
  Baseline | 16.78 (2.960) | 25.15 (9.310)
  Week 4 | 16.90 (3.539) | 22.10 (7.202)
  Week 16 | 15.60 (1.818) | 19.30 (0.245)
  Week 24 | 18.08 (2.159) | 16.63 (1.621)

14. Secondary Outcome: PRO-C3 Values Over Time: Cohort 2
Description: as for outcome 13
Time Frame: Baseline, Weeks 4, 16, 28, 40, 48
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
μg/L
  Baseline | 18.21 (3.002)
  Week 4 | 15.81 (2.948)
  Week 16 | 17.03 (2.463)
  Week 28 | 14.31 (2.362)
  Week 40 | 15.10 (2.989)
  Week 48 | 17.09 (7.967)

15. Secondary Outcome: FibroScan® Values Over Time: Cohorts 1/1b
Description: FibroScan is a type of liver elastography. Normal results are usually between 2 and 7 kilopascals (kPa), with results higher than the normal range if liver disease is present. The highest possible result is 75 kPa.
Time Frame: Baseline, Week 24
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
kPa
  Baseline | 7.28 (2.632) | 12.70 (6.988)
  Week 24 | 7.30 (3.730) | 10.55 (5.802)

16. Secondary Outcome: FibroScan® Values Over Time: Cohort 2
Description: as for outcome 15
Time Frame: Baseline, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
kPa
  Baseline | 9.89 (3.205)
  Week 48: number analyzed (Participants) | 7
  Week 48 | 8.67 (3.263)

17. Secondary Outcome: Portal Inflammation Over Time: Cohorts 1/1b
Description: Percent of participants having ≥ 1-point improvement from baseline, no change from baseline, and ≥ 1-point worsening from the baseline category in the liver biopsy parameter of portal inflammation, which was scored on a scale from 0 (none) to 3 (severe). Participants with a baseline score of 0 were not included in any of the 3 categories for this analysis.
Time Frame: Baseline, Week 24
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
percentage of participants
  ≥ 1-point improvement | 25.0 | 50.0
  no change | 50.0 | 50.0
  ≥ 1-point worsening | 25.0 | 0.0

18. Secondary Outcome: Portal Inflammation Over Time: Cohort 2
Description: as for outcome 17
Time Frame: Baseline, Week 48
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
percentage of participants
  ≥ 1-point improvement | 12.5
  no change | 37.5
  ≥ 1-point worsening | 0.0
  Baseline score = 0 | 50.0

19. Secondary Outcome: Interface Hepatitis Over Time: Cohorts 1/1b
Description: Percent of participants having ≥ 1-point improvement from baseline, no change from baseline, and ≥ 1-point worsening from the baseline category in the liver biopsy parameter of interface hepatitis, which was scored on a scale from 0 (none) to 3 (severe). Participants with a baseline score of 0 were not included in any of the 3 categories for this analysis.
Time Frame: Baseline, Week 24
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
percentage of participants
  ≥ 1-point improvement | 50.0 | 0.0
  no change | 0.0 | 100.0
  ≥ 1-point worsening | 25.0 | 0.0
  Baseline score = 0 | 25.0 | 0.0

20. Secondary Outcome: Interface Hepatitis Over Time: Cohort 2
Description: as for outcome 19
Time Frame: Baseline, Week 48
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
percentage of participants
  ≥ 1-point improvement | 25.0
  no change | 25.0
  ≥ 1-point worsening | 0.0
  Baseline score = 0 | 50.0

21. Secondary Outcome: Lobular Inflammation Over Time: Cohorts 1/1b
Description: Percent of participants having ≥ 1-point improvement from baseline, no change from baseline, and ≥ 1-point worsening from the baseline category in the liver biopsy parameter of lobular inflammation, which was scored on a scale from 0 (none) to 3 (severe). Participants with a baseline score of 0 were not included in any of the 3 categories for this analysis.
Time Frame: Baseline, Week 24
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
percentage of participants
  ≥ 1-point improvement | 0.0 | 0.0
  no change | 25.0 | 50.0
  ≥ 1-point worsening | 50.0 | 50.0
  Baseline score = 0 | 25.0 | 0.0

22. Secondary Outcome: Lobular Inflammation Over Time: Cohort 2
Description: as for outcome 21
Time Frame: Baseline, Week 48
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
percentage of participants
  ≥ 1-point improvement | 0.0
  no change | 62.5
  ≥ 1-point worsening | 12.5
  Baseline score = 0 | 25.0

23. Secondary Outcome: Hepatocyte Cell Death Over Time: Cohorts 1/1b
Description: Percent of participants having ≥ 1-point improvement from baseline, no change from baseline, and ≥ 1- point worsening from the baseline category in the liver biopsy parameter of hepatocyte cell death. Hepatocyte Cell Death Score: 0 = No acidophil bodies; 1 = Few acidophil bodies; 2 = Many acidophil. Participants with a baseline score of 0 were not included in any of the 3 categories for this analysis.
Time Frame: Baseline, Week 24
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 4 | 4
percentage of participants
  ≥ 1-point improvement | 0.0 | 0.0
  no change | 25.0 | 0.0
  ≥ 1-point worsening | 25.0 | 25.0
  Baseline score = 0 | 50.0 | 75.0

24. Secondary Outcome: Hepatocyte Cell Death Over Time: Cohort 2
Description: Percent of participants having ≥ 1-point improvement from baseline, no change from baseline, and ≥ 1-point worsening from the baseline category in the liver biopsy parameter of hepatocyte cell death. Hepatocyte Cell Death Score: 0 = No acidophil bodies; 1 = Few acidophil bodies; 2 = Many acidophil. Participants with a baseline score of 0 were not included in any of the 3 categories for this analysis.
Time Frame: Baseline, Week 48
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
percentage of participants
  ≥ 1-point improvement | 0.0
  no change | 62.5
  ≥ 1-point worsening | 0.0
  Baseline score = 0 | 37.5

25. Secondary Outcome: Meta-analysis of Histological Data in Viral Hepatitis (METAVIR) Fibrosis Stage Score Over Time: Cohorts 1/1b
Description: Percent of participants having ≥ 1-point improvement from baseline, no change from baseline, and ≥ 1- point worsening from the baseline category in the METAVIR fibrosis stage score. The METAVIR scoring system is a system used to assess the extent of inflammation and fibrosis by histopathological evaluation in a liver biopsy of patients with hepatitis C. The stage represents the amount of fibrosis or scarring. Participants with a baseline score of 0 were not included in any of the 3 categories for this analysis.
  F0: no fibrosis F1: portal fibrosis without septa F2: portal fibrosis with few septa F3: numerous septa without cirrhosis F4: cirrhosis
Time Frame: Baseline, Week 24
Population: Safety Analysis Set: all participants who received at least one dose of study drug. Participants with an assessment at the given time point.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1
Number analyzed (Participants) | 3 | 4
percentage of participants
  ≥ 1-point improvement | 0.0 | 50.0
  no change | 100.0 | 50.0
  ≥ 1-point worsening | 0.0 | 0.0

26. Secondary Outcome: Meta-analysis of Histological Data in Viral Hepatitis (METAVIR) Fibrosis Stage Score Over Time: Cohort 2
Description: as for outcome 25
Time Frame: Baseline, Week 48
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 8
percentage of participants
  ≥ 1-point improvement | 50.0
  no change | 12.5
  ≥ 1-point worsening | 25.0
  Baseline score = 0 | 12.5

27. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence which does not necessarily have to have a causal relationship with this treatment. Serious Adverse Event (SAE) is an AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, Is a congenital anomaly/birth defect, Is a medically important event or reaction. TEAEs are AEs with onset after administration of the study drug, or when a preexisting medical condition increases in severity or frequency after study drug administration. Not related events include those reported as 'Not Related' to study drug. Related events include those reported as 'Possibly Related' or 'Probably Related' to study drug.
Time Frame: From first dose of study drug up to a maximum duration of study follow-up of 202 weeks.
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1 | ARO-AAT 200 mg Cohort 2
Number analyzed (Participants) | 4 | 4 | 8
participants
  ≥ 1 TEAE | 4 | 4 | 8
  ≥ 1 Serious TEAE | 0 | 3 | 5
  TEAE Severity = Mild | 3 | 1 | 2
  TEAE Severity = Moderate | 1 | 3 | 4
  TEAE Severity = Severe | 0 | 0 | 2
  TEAE = Not Related to Study Drug (SD) | 1 | 2 | 3
  TEAE = Related to SD | 3 | 2 | 5
  TEAE Injection Site Reaction (ISR) Severity = Mild | 2 | 1 | 3
  TEAE ISR Severity = Moderate | 0 | 0 | 1
  TEAE ISR Severity = Severe | 0 | 0 | 0
  TEAE Leading to SD Discontinuation | 0 | 0 | 0
  TEAE Requiring Dose Interruption of SD | 0 | 1 | 3
  TEAE Leading to PRemature Withdrawal From Study | 0 | 0 | 0
  TEAE Causing Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For a maximum duration of study follow-up of 202 weeks.
Description: Includes SAEs from time of screening.
Arm/Group | ARO-AAT 100 mg Cohort 1b | ARO-AAT 200 mg Cohort 1 | ARO-AAT 200 mg Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 4/4 | 5/8
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARO-AAT 100 mg Cohort 1b (N=4) | ARO-AAT 200 mg Cohort 1 (N=4) | ARO-AAT 200 mg Cohort 2 (N=8)
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
Viral myocarditis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARO-AAT 100 mg Cohort 1b (N=4) | ARO-AAT 200 mg Cohort 1 (N=4) | ARO-AAT 200 mg Cohort 2 (N=8)
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 0
Dental implantation (Surgical and medical procedures) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 3
Injection site reaction (General disorders) | 1 | 0 | 2
Fatigue (General disorders) | 2 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 1
Injection site inflammation (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0
Denture wearer (Social circumstances) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Loss of libido (Psychiatric disorders) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood glucose increased (Investigations) | 0 | 1 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1
Coagulation test abnormal (Investigations) | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Spirometry abnormal (Investigations) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 2 | 0 | 1
Piriformis syndrome (Nervous system disorders) | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 6
COVID-19 (Infections and infestations) | 3 | 3 | 4
Anal candidiasis (Infections and infestations) | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Colitis (Infections and infestations) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor retains first right to publish results for this multi-center study, and thereafter can review results communications prior to release and can embargo communications regarding trial results for a period that is 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication of results but can require removal of its confidential information (excluding results).

DOCUMENTS (2):
  • Study Protocol (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03946449/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT03946449/SAP_001.pdf